CLINICAL TRIAL: NCT04181502
Title: Randomized, Single-blind Study of Remote Ischemic Preconditioning in Hepatectomies
Brief Title: Ischemic Preconditioning at a Distance in Liver Surgery
Acronym: HEPATOPROTECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2017_66; 2018-A03038-47 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-11-20; First posted 2019-11-29 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Liver Diseases
Keywords: Remote ischemic preconditioning; liver resection; liver clearance.
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inflation of a pneumatic tourniquet (Experimental)
  Interventions: Procedure: pneumatic tourniquet
- No inflation (Sham Comparator): No inflation of the pneumatic tourniquet placed on the lower limb
  Interventions: Other: No inflation

INTERVENTIONS:
Procedure: pneumatic tourniquet — a pneumatic tourniquet around 200 mmHg after venous chase of the lower limb, during 5 minutes then deflated. Repeated twice after general anaesthesia and prior to incision.
  Arms: Inflation of a pneumatic tourniquet
Other: No inflation — No inflation of the pneumatic tourniquet placed on the lower limb
  Arms: No inflation

SUMMARY:
During hepatic transection, it exists a high risk of perioperative blood loss. The haemorrhage and its consequences (hypovolemia and blood transfusion) might impact the short and long term morbidity The vascular control by hepatic pedicle clamping (Pringle's maneuver) or total hepatic vascular exclusion, helps minimizing blood loss and leads to a more extensive hepatic resection.

Side effects of vascular control result of ischemia-reperfusion injury (IRI) : these reperfusion lesions results of different mechanisms than those responsible for the ischemic one. IRI cause lesions and postoperative dysfunction of the remaining liver.

Among strategies to reduce the adverse effects of IRI : ischaemic preconditioning (IPC) has been described. It can be either mechanical (intermittent hepatic pedicle clamping) or pharmacological (sevoflurane inhalation).

Short intermittent vascular occlusions in a organ might produce a resistance to a longer ischaemic period. It is certainly a physiological organ adaptation to tissue hypoxemia, which has a therapeutic potential when targeted.

During liver resection, ischaemic preconditioning is realised with periods of hepatic pedicle clamping and unclamping. It decrease morbidity and mortality and prevent postoperative hepatocellular insufficiency due to clamping and IRI at day 5.

Ischaemic preconditioning may also be applied remotely. Indeed, it is shown that short ischaemic periods in a target organ can also have a protective effect on distant others. This mechanism involve three signalling pathways : neuronal , humoral and systemic pathways.

In a previous randomized study, Kanoria and al, demonstrated that the remote ischaemic preconditioning group has shown significant lower rates of serum transaminases and higher liver clearance (spectrophotometry method) than the control group.

A latest study, measuring postoperative prothrombin rates has shown improved liver recovery due to halogen agents such as sevoflurane.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled carcinogenic laparoscopy or laparotomy liver resection
* Insured under the social security system
* Inclined to comply to the study protocol and its duration.

Exclusion Criteria:

* Patient under guardianship
* Pregnancy or breastfeeding
* Severe lower limb vascular disease
* Emergency surgery
* Contraindication of a treatment from the protocol
* Psychological disorder with difficulty to accede the protocol
* Absence of written informed consent
* Refusal to sign the protocol
* Non-registration to the social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-06-16 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Indocyanine green clearance | at 5 days after liver resection
  Indocyanine green clearance (%/min) by indocyanine green retention, measured with Limon pulse spectrophotometry method.

SECONDARY OUTCOMES:
Serum transaminases rates | at day 1,day 3 and day 5 post-hepatectomy.
Prothrombin rate | at day 5 post-hepatectomy.
the Kidney Disease: Improving Global Outcomes (KDIGO) score | at day 1,day 3 and day 5 post-hepatectomy.
  The score varies from 1 to 4.
the Clavien & Dindo score | at day 30 post-hepatectomy
  this classification in order to rank a post operative complications. It consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V)
duration of stay in the hospital. | at day 30 post-hepatectomy

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Lebuffe, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France